CLINICAL TRIAL: NCT02763306
Title: Dermal Cryotherapy in Patients Undergoing Abdominoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-15-002
Record Dates: First submitted 2016-04-15; First posted 2016-05-05 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment with cryotherapy (Experimental): Treatment with dermal cooling system.
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Treatment with dermal cooling system.

SUMMARY:
A prospective, interventional, single-arm study to evaluate histologic changes in skin following cryotherapy with the study device.

DETAILED DESCRIPTION:
This study is to include healthy adults who intend to undergo an abdominoplasty surgery, and agree to have small areas of their middle and lower abdomen exposed to cooling with the Dermal Cooling System within 180 days before the planned surgery. Exposure of multiple test sites will be completed in areas of skin that will be excised as part of the abdominoplasty procedure. Clinical assessments of the treatment sites at 1-week post-treatment and at 1-month post-treatment intervals throughout the time period prior to surgical excision, and histologic evaluation of the treated skin will be conducted to assess skin changes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subjects eligible, consented, and scheduled for abdominoplasty.
3. Subject is willing to use photoprotection (e.g., sun avoidance) of the treated areas during the duration of the follow-up period.
4. Subject has read and signed a written informed consent form. -

Exclusion Criteria:

1. Subject has medical or surgical treatment in the area of intended treatment in the previous 6 months (e.g., liposuction, mesotherapy, hydroquinone, corticosteroids, laser surgery).
2. Subject has a known history of subcutaneous injections into the abdomen within the past six months (e.g., insulin, Enbrel).
3. Subject has a known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease).
4. Subject is taking methylxanthines (phosphodiesterase-inhibitors like amino- or theophylline)
5. Artificial tanning in the area of intended treatment within 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period.
6. Subject is unable or unwilling to comply with the study requirements.
7. Subject has any dermatological conditions or scars (other than stretch marks) within the area of planned abdominoplasty excision that may interfere with the ability to obtain test sites for treatment or evaluation.
8. Subject has a history of abnormal wound healing or abnormal scarring.
9. Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
10. Patient is pregnant or intending to become pregnant within the next 6 months.
11. Patient is lactating or has been lactating in the past 9 months.
12. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Histologic evaluation of treated skin | 1-180 days
  Identify a range of treatment parameters which elicits a response in melanocytes based upon histologic assessments.

SECONDARY OUTCOMES:
Access device or procedure-related adverse events | 1 - 180 days
  Assess adverse events and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: David Kaufman, MD, Principal Investigator — Kaufman Plastic Surgery
Locations (2):
- United States (2):
  - Kaufman Plastic Surgery, Folsom, California
  - Fremont Plastic Surgery, Fremont, California

IPD SHARING:
Plan to Share IPD: No